CLINICAL TRIAL: NCT04110808
Title: Comparative Effect of Hypotensive Anaesthesia Using Nitroglycerine vs Phentolamine on Event Related Potentials, Quantitative Electroencephalograghy and Cognitive Function in Patients Undergoing Septoplasty
Brief Title: Comparative Effect of Hypotensive Anaesthesia on Event Related Potentials, Quantitative Electroencephalograghy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mona Hussein, Neurology lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: hypotensive anaesthesia
Record Dates: First submitted 2019-09-06; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Effect of Drugs

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitroglycerine (Active Comparator): Patients will receive hypotensive anesthesia with nitroglycerine infusion via syringe pump by adding 5mg (5ml) of Nitroglycerin to 45ml of normal saline making it to final concentration of 100μg/ml at the rate of 0.5- 10 μg/kg/min according to the patients desired target blood pressure.
  Interventions: Drug: hypotensive anaesthesia using Nitroglycerine
- Phentolamine (Other): Patients will receive hypotensive anesthesia with phentolamine infusion via syringe pump by adding 20 mg (2ml) of Phentolamine to 48 ml of normal saline making it to final concentration of 0.4 mg/ml at the rate of 0.1-2 mg/min according to the patients desired target blood pressure.
  Interventions: Drug: hypotensive anaesthesia using Nitroglycerine

INTERVENTIONS:
Drug: hypotensive anaesthesia using Nitroglycerine — effect of hypotensive anaesthesia using Nitroglycerine vs Phentolamine on Event related potentials, quantitative Electroencephalograghy and cognitive function
  Phentolamine group (30 patients): Patients will receive hypotensive anesthesia with phentolamine infusion via syringe pump by adding 20 mg (2ml) of Phentolamine to 48 ml of normal saline making it to final concentration of 0.4 mg/ml at the rate of 0.1-2 mg/min according to the patients desired target blood pressure.
  Nitroglycerine group (30 patients): Patients will receive hypotensive anesthesia with nitroglycerine infusion via syringe pump by adding 5mg (5ml) of Nitroglycerin to 45ml of normal saline making it to final concentration of 100μg/ml at the rate of 0.5- 10 μg/kg/min according to the patients desired target blood pressure.
  Other Names: hypotensive anaesthesia using Phentolamine

SUMMARY:
AIM OF THE WORK The aim of this work was to compare the effect of hypotensive anaesthesia using Nitroglycerine versus phentolamine on Event related potentials, quantitative Electroencephalograghy and cognitive function, in patients undergoing septoplasty.

DETAILED DESCRIPTION:
METHODS:

Study design and population: This is a pilot prospective randomized clinical trial that will be carried out on 60 patients candidate for septoplasty subjected to general hypotensive anaesthesia. The patients will be recruited from Ear, nose and throat surgery department, Beni-Suef University Hospital. All the participants will be required to offer a written informed consent

Sampling Technique:

Patients will be randomly assigned into one of two equal groups; the first group will receive nitroglycerine (30 participants) (nitroglycerine group) and the second group will receive phentolamine (30 participants) (phentolamine group). Randomization will be carried out using a closed opaque envelope technique with the anesthetist will pick up a sealed envelope which contains a paper with the name of the group to which the patient will be randomized is written. Whichever the group written on the paper, the patient will be scheduled to it.

All included patients will be subjected to the following:

1) Cognitive assessment:

Cognitive functions for the patients will be assessed (preoperative and 1 week postoperative) using the following psychometric tests:

1. Paired Associate Learning test (PALT) Aim: to assess auditory verbal memory. The test uses the concept of semantic cueing

   .
2. Benton Visual Retention test (BVRT) Aim: to assess visual perceptual, visual memory, visual motor and visuoconstructive abilities.

2) Neurophysiological assessment: Digital Electroencephalograghy (EEG), quantitative Electroencephalograghy (QEEG) and Event related potentials (ERPs) and will be done for all included patients (preoperative and 1 week postoperative).

Statistical analysis The sample size will be calculated using G*Power version 3.1.9.2 Software based on this pilot study. The probability of type I error (α) will be 5%, and the statistical power (1-β) should exceed 80%. The data will be coded and entered using: the statistical package for social science version 15 (SPSS v 15). Descriptive statistics will be reported as mean ± SD and number (%) for categorical variables. Student t- test will be used for comparison between means of two unpaired groups of quantitative variables. Paired sample t- test will be used for comparison between means of two paired groups of quantitative variables. Chi square test will be used for comparison between two groups of categorical data. Mixed ANOVA test will be used for comparing paired data in two unpaired groups. The probability/significance value (P value) ≥ 0.05 is not statistically significant and <0.05 is statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidate for septoplasty
* Patients from both sexes, aged between 20-50 years

Exclusion Criteria:

* Patients who develop intraoperative shock or major bleeding
* Patients with ischemic heart diseases, heart block, congestive heart failure, valvular heart diseases, or uncontrolled hypertension
* Patients with a history of central neurological system disorder
* Patients with concomitant medical or metabolic illness known to affect cognition
* Pregnant females
* Allergy to any of the anaesthetic or hypotensive drugs used in the study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Paired Associate Learning test for assessment of Cognitive function | 1 week
  Comparative effect of hypotensive anaesthesia using Nitroglycerine vs Phentolamine
Benton Visual Retention test for assessment of Cognitive function | 1 week
  Comparative effect of hypotensive anaesthesia using Nitroglycerine vs Phentolamine

SECONDARY OUTCOMES:
Quantitative Electroencephalograghy for assessment of electrical activity of the brain | 1 week
  Comparative effect of hypotensive anaesthesia using Nitroglycerine vs Phentolamine
Event related potentials (ERP ) P300 for neurophysiological assessment of cognition | 1 week
  Comparative effect of hypotensive anaesthesia using Nitroglycerine vs Phentolamine